CLINICAL TRIAL: NCT03687554
Title: A Phase I, Single-Center, Open-label, Single Dose Pharmacokinetic and Tolerability Study of GZ402671 in Subjects With Mild, Moderate and Severe Renal Impairment, and in Matched Subjects With Normal Renal Function
Brief Title: Effect of Venglustat in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POP14499; U1111-1205-3215 (Other: UTN)
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers; Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — venglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venglustat (Experimental): Single dose of Venglustat is given, orally under fasting conditions
  Interventions: Drug: Venglustat GZ/SAR402671

INTERVENTIONS:
Drug: Venglustat GZ/SAR402671 — Pharmaceutical form: Hard Capsule Route of administration: Oral

SUMMARY:
Primary Objective:

To study the effect of mild, moderate and severe renal impairment on the pharmacokinetics (PK) of Venglustat following a single dose.

Secondary Objective:

To assess the tolerability of Venglustat given as a single dose in subjects with mild, moderate and severe renal impairment in comparison with matched subjects with normal renal function.

DETAILED DESCRIPTION:
Approximately 41 days, including a 21-day screening period, a 1-day treatment period, followed by a 9-day period of plasma sampling for assessment of primary endpoints.

ELIGIBILITY:
Inclusion criteria:

For all Subjects:

* Male and/or female subjects, between 18 and 79 years of age, inclusive.
* Body weight between 50.0 and 115.0 kg, inclusive, if male, and between 40.0 and 100.0 kg, inclusive, if female, body mass index between 18.0 and 34.9 kg/m2, inclusive
* Normal electrocardiogram (ECG)
* Having given written informed consent prior to undertaking any study-related procedure
* Not under any administrative or legal supervision
* Male subject, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method according to the following algorithm: (condom) plus (spermicide or intra-uterine device or hormonal contraceptive) from the inclusion up to 4 months after the last dosing
* Male subject, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 4 months after the last dosing
* Male subject has agreed not to donate sperm from the inclusion up to 4 months after the last dosing
* Female subject must use a double contraception method including a highly effective method of birth control from at least 30 days prior to the inclusion to 30 days after the last IMP administration, except if she has undergone sterilization (documented) at least 3 months earlier or is postmenopausal

Specific for subjects with renal impairment:

* Stable chronic renal impairment
* Vital signs and laboratory parameters within acceptable range for subjects with renal impairment

Specific for matched healthy subjects:

* Normal renal function
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical exam)
* Normal vital signs and laboratory parameters

Exclusion criteria:

* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month)
* Blood donation, any volume, within 2 months before inclusion
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension judged clinically relevant by the Investigator
* Any significant change in chronic treatment medication within 14 days before inclusion
* Any drug which could impact by any mechanism of action, the pharmacokinetics of the investigational medicinal product, including moderate and strong cytochrome P3A (CYP3A) inhibitors or inducers; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab)
* Positive result on urine drug screen or plasma alcohol test
* Active hepatitis, hepatic insufficiency
* If female, pregnancy [defined as positive β-Human Chorionic Gonadotropin (β-HCG) blood test], breast-feeding

Specific for subjects with renal impairment:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastrointestinal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness
* Acute renal failure (de novo or superimposed on preexisting chronic renal impairment), nephrotic syndrome
* History of or current hematuria of urologic origin that limits the subject's participation in the study
* Subjects requiring dialysis during the study

Specific for matched healthy controls:

- Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female) or infectious disease, or signs of acute illness

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameters of Venglustat: Area under the curve (AUC) | Day 1 to Day 10
  Venglustat area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
Venglustat plasma pharmacokinetic (PK) parameter: Cmax | Day 1
  Maximum plasma concentration observed (Cmax)
Venglustat plasma pharmacokinetic (PK) parameter: AUClast | Day 1 to Day 10
  Area under the plasma concentration versus time curve calculated from time zero to the real time tlast (AUClast)
Venglustat plasma pharmacokinetic (PK) parameter: unbound Cmax | Day 1 to Day 10
  Maximum plasma concentration observed of unbound drug (unbound Cmax)
Venglustat plasma pharmacokinetic (PK) parameter: unbound AUC | Day 1 to Day 10
  Change in unbound Venglustat area under the plasma concentration versus time curve (unbound AUC)
Venglustat plasma pharmacokinetic (PK) parameter: CL/F | Day 1 to Day 10
  Apparent total body clearance of Venglustat from plasma (CL/F)
Venglustat plasma pharmacokinetic (PK) parameter: Vss/F | Day 1 to Day 10
  Apparent volume of distribution of Venglustat at steady state (Vss/F)
Venglustat plasma pharmacokinetic (PK) parameter: fu | Day 1 to Day 10
  Fraction of unbound venglustat in plasma (fu)
Venglustat plasma pharmacokinetic (PK) parameter: t1/2z | Day 1 to Day 10
  Terminal half-life associated with the terminal slope (t1/2z)
Venglustat plasma pharmacokinetic (PK) parameter: t1/2eff | Day 1 to Day 10
  Effective half-life (t1/2eff)
Venglustat urine pharmacokinetic (PK) parameter: Ae(0-24) | Day 1 and Day 2
  Cumulated amount excreted in urine from time 0 to time 24h after Venglustat administration
Venglustat urine pharmacokinetic (PK) parameter: fe(0-24) | Day 1 and Day 2
  Fraction of dose excreted in urine from time 0 to time 24h after Venglustat administration
Venglustat urine pharmacokinetic (PK) parameter: CLR(0-24) | Day 1 and Day 2
  Renal clearance of the drug determined in the 0-24h interval (CLR(0-24))
Venglustat plasma pharmacokinetic (PK) parameter: Rac,pred | Day 1 to Day 10
  Predicted accumulation ratio (Rac,pred)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 8400001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org